CLINICAL TRIAL: NCT02207348
Title: A Randomised, Open-label, Single-centre, Two-period, Cross-over Trial Investigating Bioequivalence Between Single-dose Liraglutide Administered Subcutaneously With Two Different Pen-injectors
Brief Title: Investigating Bioequivalence Between Single-dose Liraglutide Administered Subcutaneously With Two Different Pen-injectors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN8022-4162; 2014-000216-34 (EudraCT Number); U1111-1152-1391 (Other: WHO)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide 0.6 mg s.c. with FlexPen® (Experimental)
  Interventions: Drug: liraglutide
- Liraglutide 0.6 mg s.c. with the PDS290 pen-injector (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Each subject will receive two single doses of 0.6 mg liraglutide (one with each of the two pen-injectors)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate bioequivalence between single-dose liraglutide administered subcutaneously with two different pen-injectors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-60 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) greater than or equal to 27.0 and less than 35.0 kg/m^2
* Bodyweight up to 130.0 kg (inclusive)
* HbA1c (glycosylated haemoglobin) below 6.5%

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices), or sexual abstinence or vasectomised partner
* History or presence of cancer, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrine (incl. diabetes), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders that might have impact on the trial, as judged by the investigator
* Use of any prescription or non-prescription medication, except for paracetamol, acetylsalicylic acid, contraceptives and vitamins (but including mega-dose vitamin therapy, as judged by the investigator) within 2 weeks before the trial defined as screening
* Significant history of alcoholism or drug/chemical abuse within 1 year from screening, or a positive result of the urine drug screen or alcohol breath test, or consuming more than 21 units of alcohol per week (one unit of alcohol equals about 250 mL of beer or lager, one glass of wine (120 mL), or 20 mL spirits)
* Smoking more than 5 cigarettes, or the equivalent, per day and unable to refrain from smoking during the in-house periods

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under the liraglutide plasma concentration time curve from 0 to last quantifiable observation (tz) after single dose | 0-72 hours following administration of 0.6 mg liraglutide
Maximum observed liraglutide plasma concentration after single dose | 0-72 hours following administration of 0.6 mg liraglutide

SECONDARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From baseline to follow-up (up to 3 weeks). Baseline is defined as time of first trial drug administration at Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com